CLINICAL TRIAL: NCT01577030
Title: Hypotensive Effects of Conventional Dairy Products: Role of Arterial Stiffness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: LH002
Record Dates: First submitted 2012-04-10; First posted 2012-04-13 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Prehypertension; Stage-1 Hypertension
MeSH Terms: conditions — Prehypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dairy (Experimental): Add 4 daily servings of non-fat dairy to diet for a period of 4 weeks
  Interventions: Dietary Supplement: Non-fat dairy
- Fruit (Active Comparator): Add 4 daily servings of fruit to diet, remove all dairy from diet for a period of 4 weeks
  Interventions: Dietary Supplement: Add 4 servings fruit

INTERVENTIONS:
Dietary Supplement: Non-fat dairy — Add 4 daily servings per day of non-fat dairy (yogurt, milk, cheese) for a period of 4 weeks
  Arms: Dairy
Dietary Supplement: Add 4 servings fruit — Add 4 daily servings of fruit (fruit cup, apple sauce, orange juice) and remove all dairy for a period for 4 weeks
  Arms: Fruit

SUMMARY:
Elevated systolic blood pressure is by far the largest single contributor to cardiovascular risks in middle-aged and older adults. Lifestyle modifications, including dietary modifications, are the first line approach for treating and preventing hypertension. The general aim of the proposed study is to address the efficacy of conventional dairy products as part of the normal routine diet for lowing arterial blood pressure in middle-aged and older adults with elevated blood pressure. The investigators hypothesize that the dietary intervention including dairy products will induce significant decreases in arterial blood pressure in this population. A secondary aim will be to test the hypothesis that these reductions in systolic blood pressure will be associated with increases in arterial stiffness/compliance and endothelial vasodilatory function.

ELIGIBILITY:
Inclusion Criteria:

* Prehypertension or stage-1 hypertension

Exclusion Criteria:

* Consume > 3 servings of dairy or fruit per day
* Strenuous physical activity > 3 time per week
* Lactose intolerance, pregnancy, lactation, and/or alcohol abuse
* Taking cardiovascular-acting drugs
* Overt cardiovascular disease, metabolic disease, GI disorders and/or renal disease

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-01; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Seated blood pressure | 4 weeks

SECONDARY OUTCOMES:
24-hour ambulatory blood pressure | 4 weeks
Carotid arterial compliance | 4 weeks
Arterial stiffness | 4 weeks
Flow mediated dilation | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hirofumi Tanaka, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- The University of Texas at Austin, Cardiovascular Aging Research Laboratory, Austin, Texas, United States

REFERENCES:
- [Derived] Machin DR, Park W, Alkatan M, Mouton M, Tanaka H. Effects of non-fat dairy products added to the routine diet on vascular function: a randomized controlled crossover trial. Nutr Metab Cardiovasc Dis. 2015 Apr;25(4):364-9. doi: 10.1016/j.numecd.2015.01.005. Epub 2015 Jan 31. PMID 25770758
- [Derived] Machin DR, Park W, Alkatan M, Mouton M, Tanaka H. Hypotensive effects of solitary addition of conventional nonfat dairy products to the routine diet: a randomized controlled trial. Am J Clin Nutr. 2014 Jul;100(1):80-7. doi: 10.3945/ajcn.114.085761. Epub 2014 May 7. PMID 24808486